CLINICAL TRIAL: NCT05046288
Title: A 3-month Cycle of Weekly Montreal Museum of Fine Arts Guided Tours Oto Promote Social Inclusion, Well-being, Quality of Life and Health in Older Community Members Experiencing Social Isolation
Brief Title: Virtual Guided Tour of the MMFA for Prevention of Social Isolation
Acronym: VGV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Senior researcher, Director of laboratory, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-1338
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Social Isolation; Well Aging; Quality of Life; Healthy Aging
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants will participate to the 3-month cycle of virtual guided tour of the MMFA and will complete assessments at M0 and at M3
  Interventions: Other: Virtual guided tours
- Group 2 (No Intervention): Participants will not participate to the 3-month cycle of virtual guided tour of the MMFA but will complete assessments at M0 and at M3

INTERVENTIONS:
Other: Virtual guided tours — The intervention is a participatory art-based activity which consists in MMFA virtual guided tours. Each virtual guided tour is performed with a group of 6 to 7 participants. They meet online one time per week for a 30 to 45 min of a guided tour during a 3-month period. Each tour is different and supervised by a MMFA trained guide.
  Arms: Group 1

SUMMARY:
It has previously been reported that participatory art-based activities may improve social inclusion, well-being, quality of life and health condition. Findings from the investigator's first study seem to confirm that the MMFA participatory art-based activity may improve well-being, quality of life and health condition in older community dwellers. However, these studies were performed before the COVID-19 crisis and were guided tours performed at the MMFA. A pilot study on virtual guided tour has been performed during COVID-19 pandemic (spring 2021). There is a need to confirm benefits with a randomized clinical trial.

The hypothesize for this study is that a 3-month cycle of virtual weekly MMFA tours may induce changes in social isolation, well-being, quality of life and health condition (i.e., reduction of frailty) in older community dwellers. Because there is a positive correlation between severity of frailty and the occurrence of undesirable events like Emergency department (ED) visits and hospitalizations, the investigator hypothesizes that virtual guided tours may decrease the frequency of ED visits and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* age 65 and over;
* having a low level of social inclusion defined with the 11-item Duke Social Support Index (DSSI) score ≤ 26/3323;
* living in Quebec, at home in an urban area;
* reading, understanding and writing the languages of the recruitment centre (i.e., French or English or Chinese mandarin) because all the questionnaires are available in French, in English and in Chinese mandarin, and because the guides of the museum performing the virtual guided tours speak French and/or English, with a translator in Chinese mandarin.
* Having an Internet access and an electronic device (smartphone, laptop, computer and/or tablet with a functional cam) at the participant's place of living as the repetitive assessments for this study will be performed on the web platform of the CRIUGM, and the guided tours will be virtual.

Exclusion Criteria:

* Cannot participate to a clinical trial at the same time, to avoid interferences with the outcomes of the studied intervention in this protocol.
* Having participated to a participatory art-based activity of the MMFA during the 3 month-period before the recruitment. A participation to any other museum activities may be assimilate to an intervention. As it could interfere with our outcomes, participants are not allowed to participate to any other museum activity, in any museum, during their 3-month participation. We previously showed that museum activities may change the outcomes studied in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Social isolation | 3 months
  social isolation which will be assessed using the 11-item Duke Social Support Index (DSSI). .The index comprises two subscales: social interaction (i.e., frequency of interactions) and subjective support (i.e., satisfaction with emotional support provided). DSSI score ranges from 11 to 33, increased score indicating higher levels of social insertion. The scores of the 11 items are combined and categorized as low-fair (score ≤26), high (score 27-29) and very high (score 30-33). We will use as primary outcome the mean score of 11-item DSSI and its distribution in three categories.

SECONDARY OUTCOMES:
Frailty | 3 months
  The frailty which will be assessed using the CRIUGM Self-AdMinistered questionnaire (CESAM).
  The CESAM is composed of a maximum of 28 items exploring age, sex, nutrition, place of life, social resources, number of drugs taken on a daily basis, memory complaint, mood and general feeling, fatigue, activities of daily living scale, instrumental activities of daily living scale, physical activity and history of previous falls. Items correspond to a question in closed-ended format (i.e., yes or no, or calling for a specific answer). The CESAM provides two complementary information: 1) A global score of frailty ranged from 0 (i.e., best health and functional condition) to 18 (i.e., worse health and functional condition) and 2) Categorized health condition in four levels (vigorous with a score between 0 and 3, mild frailty with a score between 4 and 7, moderate frailty with a score bet
socio-geriatric vulnerability | 3 months
  socio-geriatric vulnerability will be assessed using the digital form of a self-administered questionnaire ESOGER. The ESOGER is composed of a maximum of 15 questions exploring the COVID risk, the COVID past history, COVID vaccination the social isolation risk due to COVID (access to food, home support and healthcare, contact with external persons, anxiety). Items correspond to a question in closed-ended format (i.e., yes or no, or calling for a specific answer). Incident planned and unplanned visits to physicians, Emergency Department (ED) and hospitalization during the 3-month cycle of virtual weekly MMFA tours will be only recorded at the end of the cycle.
Well-being | 3 months
  Well-being will be assessed using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) self-questionnaire. WEMWBS is a validated questionnaire composed by 14 positively worded item scale with five response categories. It covers most aspects of positive mental health (positive thoughts and feelings).
quality of life | 3 months
  quality of life will be assessed using the EuroQol-5D (EQ-5D). This test is a standardized measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. It provides a simple descriptive profile and a single index value for health status.
  EQ-5D is composed of two parts:
  * a questionnaire of five questions with score per question ranged from 1 (i.e., no issue) to 5 (i.e., worse issue),
  * and a visual analogic scale of how good or bad participant health was. This scale is numbered from 0 (i.e., worse health participant can imagine) to 100 (i.e., best health participant can imagine).
compliance | 3 months
  compliance to the MMFA visits will be assessed by counting the number of virtual tours completed during the 3-month period of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beauchet O, Matskiv J, Galery K, Goossens L, Lafontaine C, Sawchuk K. Benefits of a 3-month cycle of weekly virtual museum tours in community dwelling older adults: Results of a randomized controlled trial. Front Med (Lausanne). 2022 Aug 16;9:969122. doi: 10.3389/fmed.2022.969122. eCollection 2022. PMID 36052331